CLINICAL TRIAL: NCT01914250
Title: Pain Associated With Neonatal Frenotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 01 Dated 01 August 2012
Record Dates: First submitted 2013-07-17; First posted 2013-08-02 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Pain
Keywords: Frenotomy; Pain
MeSH Terms: conditions — Pain

ARMS (1):
- 2 (Active Comparator): Topical Anesthetic, 2% Tetracaine oral gel - Group A Topical Anesthetic, 20% Benzocaine oral gel - Group B
  Interventions: Drug: Analgesic effect of topical tetracaine 2 %

INTERVENTIONS:
Drug: Analgesic effect of topical tetracaine 2 % — The patient will be held by the parents and comforted after local anesthesia is applied by a research investigator. Then, he will be placed on procedure's board repositioned for clipping, restrained by the parent/nurse (holding both head and arms, keeping with conventional practice). Exactly 5 minutes after the topical anesthetic was applied, the pediatric dentist will press down the chin gently straddling the frenulum while and holding it in place with visualization of tongue base. Then the frenulum will be snipped along the underside of the tongue to its base. The area will be checked to ensure complete release. Bleeding will be controlled by pressuring with a 2x2 gauze pad under the tongue. A study investigator will film the procedure using GO PRO Video Camera mounted on the forehead of the pediatric dentist

SUMMARY:
The present study sought to examine the efficacy of two oral anesthetic drugs in reducing the pain associated with neonatal frenotomy.

ELIGIBILITY:
Inclusion Criteria:

infants diagnosed with ankyloglossia at the nursery of the RHCC, who will be referred by a qualified neonatologist to the OCAD for a routine tongue-tie frenotomy procedure because of breast feeding difficulties.

* Ankyloglossia type 1 or 2 Exclusion criteria
* Abnormal oral or nasopharyngeal anatomy
* Any known congenital malformations
* Ankyloglossia type 3 or 4

Exclusion Criteria:

-

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Neonatal Facial Coding System (NFCS) | During procesure

SECONDARY OUTCOMES:
Cry Duration | Post procedure

OTHER OUTCOMES:
Visual Analog Score (VAS) | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dror - Aizenbud, Professor, Principal Investigator — Chairman Craniofecial Department, Rambam Medical Center
Locations (1):
- Rambam HealthCare Campus, Haifa, Israel

REFERENCES:
- [Derived] Shavit I, Peri-Front Y, Rosen-Walther A, Grunau RE, Neuman G, Nachmani O, Koren G, Aizenbud D. A Randomized Trial to Evaluate the Effect of Two Topical Anesthetics on Pain Response During Frenotomy in Young Infants. Pain Med. 2017 Feb 1;18(2):356-362. doi: 10.1093/pm/pnw097. PMID 28204733